CLINICAL TRIAL: NCT06739720
Title: A Randomized, Waitlist-controlled Clinical Study on the Efficacy and Safety of Lingzhi-containing Dietary Supplement CP003 on Chronic Fatigue and Post-COVID Fatigue
Brief Title: RCT of Efficacy and Safety of CP003 on CFS/ME or Post-COVID Fatigue
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Innovation and Technology Commission, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKWC-2024-320
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Chronic Fatigue Syndrome (CFS); Post-COVID ME/CFS
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to either the intervention group or the waitlist group. The intervention group receives CP003 capsules (5 capsules once daily) for 6 weeks. The waitlist group undergoes a 6-week waiting period without any treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receive CP003 capsules (5 capsules once daily) for 6 weeks, followed by a 6-week follow-up period.
  Interventions: Drug: LingZhi capsule
- Waitlist group (No Intervention): Participants initially wait for 6 weeks after randomization without intervention. After the waiting period, they receive the same CP003 supplement regimen (5 capsules once daily) for 6 weeks, followed by a 6-week follow-up period.

INTERVENTIONS:
Drug: LingZhi capsule — Lingzhi-containg capsules (CP003) is a Chinese Medicine nutritional supplement manufactured by Chinese Pharm CO LTD containing: wild red ganoderma extract, ganoderma spore powder (99.9% broken wall), β-nicotinamide mononucleotide (NMN), wild yellow ganoderma extract, wild green ganoderma extract, wild purple ganoderma extract, wild white ganoderma extract, wild black sesame extract
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to test if a Lingzhi supplement (CP003) helps people with chronic fatigue or post-COVID fatigue feel better. It will also check if the supplement is safe to use. The main questions it aims to answer are:

Does the Lingzhi supplement reduce fatigue symptoms? Is it safe to take? How does it affect the body's immune system and inflammation?

Researchers will compare people taking the Lingzhi supplement to those who don't take anything (waitlist group) to see if it works.

Participants will:

* Take 5 capsules once daily for 6 weeks (or wait to start treatment if in waitlist group)
* Visit the clinic 2 times for blood tests (before and after taking the supplement)
* Complete questionnaires 3 times about their fatigue and quality of life (4 times questionnaires for waitlist group)

ELIGIBILITY:
Inclusion Criteria:

* Meet the Fukuda diagnostic definition of CFS/ME or have persisting fatigue after the infection of SARS-CoV-2
* Are able to complete a 6-week course of intervention;
* Able to complete the online validated fatigue surveys.

Exclusion Criteria:

* Have participated in any type of complements or herbal medicine within the past six months;
* Have serious medical conditions that might limit their participation in this intervention;
* Diagnosed with acute inflammation;
* Are pregnant or are planning a pregnancy in the next 3 months.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference in Chalder Fatigue Score | From baseline to 6 weeks

SECONDARY OUTCOMES:
Mean difference in Chalder Fatigue Score | From baseline to 12 weeks
Mean difference in 36-Item Short-Form Health Survey | from baseline to 6 week and 12 week
Mean difference in Fatigue Severity Score | from baseline to 6 week and 12 week
mean difference in (PROMIS) Short Form Fatigue 7A survey | from baseline to 6 week and 12 week
Mean difference in hospital anxiety and depression scale | from baseline to 6 week and 12 week
Mean difference in Pittsburgh sleep quality index | from baseline to 6 week and 12 week visit.

OTHER OUTCOMES:
Change in serum markers | From baseline to 6 weeks
  for inflammation, immunity and oxidative aging

CONTACTS AND LOCATIONS:
Locations (1):
- Specialist Clinical Centre for Teaching and Research, School of Chinese Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Xun Y, Fong TL, Chen G, Feng Y, Chan L, Wang N. Effectiveness and Safety of a Supplement Containing a Pharmacologically Active Basidiomycete Mushroom for Chronic Fatigue and Post-COVID-19 Fatigue Syndrome: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2026 Jan 20;15:e82633. doi: 10.2196/82633. PMID 41558017